CLINICAL TRIAL: NCT07394556
Title: Prospective Research on the Intervention of Myoless2.0 in Europe (PRIME)
Acronym: PRIME
Status: Not yet recruiting | Type: Observational
Sponsor: Indizen Optical Technologies, S.L.U. (Industry)
Collaborators: Hospital San Carlos, Madrid (Other); University of Minho (Other); University of Ulster (Other)
Responsible Party: Sponsor
Other Study IDs: IOT-PRIME-2026-01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Myopia Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: myopia control lens — Evaluation of the efficacy in decreasing myopia progression of the proposed ophthalmic lens prototypes.

SUMMARY:
The Goal of the study is to evaluate the rate of myopia progression with open ring myopia control spectacle lens designs compared to a commercial peripheral plus myopia control spectacle lens (CML) in European children with myopia. This is a prospective, randomized, bilateral wear, double masked, cross-over clinical trial. There will be a total of 180 participants randomized into three groups, Group 1 - 60 participants will wear the commercial peripheral plus myopia control lens (CML).

Group 2 - 60 participants will wear the Open Ring 1 (OR1) lens design. Group 3 - 60 participants will wear the Open Ring 2 (OR2) lens design. For each group, an equal balance of gender will be recruited and 50% of children will be aged between 6- 9 years old and 50% aged 10-12 years old. All groups will be required to wear spectacles for all waking hours for 12 months. After 12 months, the control group will continue wearing CML for a further 12 months; the Group 2 participants will continue wearing the OR1 lens for a further 12 months. The Group 3 participants will wear OR2 or OR3 (a modified design of OR2) based on their risk of myopia progression for a further 12 months

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 6 to 12 completed years (6 and 12 years inclusive), irrespective of gender.
* For each group, an equal balance of gender will be recruited and 50% of children will be aged between 6- 9 years old and 50% aged 10-12 years old.
* Be cycloplegic autorefraction spherical component -0.50 D to -6.00D, cylinder no more than -2.00D, and with a spherical equivalent greater than or equal to -6.00D.
* Be accompanied by parents/guardians who can read and comprehend give informed consent as demonstrated by signing a record of informed consent.
* Be willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator.
* Have ocular health findings considered to be "normal".
* Be correctable to at least 6/9.5 (20/30) or better in each eye with spectacles.
* Be willing to wear the spectacles provided by the investigators for all waking hours.

Exclusion Criteria:

* A known allergy to, or a history of intolerance to cyclopentolate or topical anesthetics.
* Had strabismus and/or amblyopia.
* Cylinder more than -2.00D
* Anisometropia greater than 1.50D spherical equivalent
* Had previous eye surgery (including strabismus surgery).
* Any ocular, systemic or other condition or disease with possible associations with myopia or affecting refractive development e.g. Marfan syndrome, retinopathy of prematurity, diabetes.
* Had any ocular injury or condition (including keratoconus and herpes keratitis) of the cornea, conjunctiva or eyelids.
* Current orthoptic treatment or vision training.
* Any anatomical, skin or other condition that would impact on the wearing of spectacles.
* Use of or need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Currently enrolled in another clinical trial.
* No previous myopia management intervention or treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Children aged between 6-12 years old from Spain, Portugal and the United Kingdom
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Myopic progression in one year | At baseline, 3, 6, 12, 18 and 24 months
  This is expressed as the change in spherical equivalent refractive state from baseline levels. Spherical equivalent refraction will be taken as the mean of the spherical equivalent refraction of five, reliable, cycloplegic autorefraction measurements on each eye with a precision of 0.12D. Myopia progression is also expressed as the change in axial length from baseline levels. Myopia progression is characterized by ocular anatomical changes, the most notable being increased axial length.

CONTACTS AND LOCATIONS:
Locations (3):
- Universidade Do Minho, Braga, Portugal
- Hospital Universitario Clínico San Carlos, Madrid, Spain
- Ulster University, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Perez C, Sanchez-Tena MA, Cleva JM, Villa-Collar C, Alvarez M, Chamorro E, Alvarez-Peregrina C. Efficacy of Asymmetric Myopic Peripheral Defocus Lenses in Spanish Children: 24-Month Randomized Clinical Trial Results. Children (Basel). 2025 Feb 6;12(2):191. doi: 10.3390/children12020191. PMID 40003293
- [Background] Sanchez-Tena MA, Cleva JM, Villa-Collar C, Alvarez M, Ruiz-Pomeda A, Martinez-Perez C, Andreu-Vazquez C, Chamorro E, Alvarez-Peregrina C. Effectiveness of a Spectacle Lens with a Specific Asymmetric Myopic Peripheral Defocus: 12-Month Results in a Spanish Population. Children (Basel). 2024 Feb 1;11(2):177. doi: 10.3390/children11020177. PMID 38397289